CLINICAL TRIAL: NCT04355494
Title: SOLIRIS® (Eculizumab) for the Treatment of Participants With Coronavirus Disease 2019 (COVID 19) - An Expanded Access Program for Hospital-based Emergency Treatment
Brief Title: SOLIRIS® (Eculizumab) Treatment of Participants With COVID-19
Status: No longer available | Type: Expanded Access
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ECU-COV-401
Record Dates: First submitted 2020-04-17; First posted 2020-04-21 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: COVID-19; Pneumonia, Viral; Acute Lung Injury/Acute Respiratory Distress Syndrome (ARDS)
Keywords: acute lung injury; acute respiratory distress syndrome; antibodies, monoclonal, humanized; complement inhibition; COVID-19; eculizumab; emergency treatment; expanded access program; hospitalization; pneumonia; severe acute respiratory syndrome; severe acute respiratory syndrome coronavirus 2; severe pneumonia; Soliris; viral
MeSH Terms: conditions — COVID-19; Pneumonia, Viral; Acute Lung Injury; Respiratory Distress Syndrome; Pneumonia; Severe Acute Respiratory Syndrome | interventions — eculizumab

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Biological: eculizumab — Eculizumab at doses of 900-1200 mg will be administered intravenously (up to 7 doses)
  Other Names: Soliris

SUMMARY:
This protocol provides access to eculizumab treatment for participants with severe COVID-19.

DETAILED DESCRIPTION:
This is an open label, multicenter, Expanded Access Program (EAP) to allow participants with a confirmed diagnosis of SARS-CoV-2 infection, and a clinical presentation consistent with COVID-19 severe pneumonia, acute lung injury, or ARDS to be treated with eculizumab. Participants admitted to a designated hospital facility who qualify for emergency treatment will be administered eculizumab up to 7 times during their treatment course (5 mandatory doses and up to 2 optional doses, per Investigator assessment).

The EAP consists of a Screening Period of up to 7 days, a 4-week Treatment Period, a final in-hospital assessment on Day 29 or day of discharge, whichever occurs first, and 3 monthly safety follow up visits (to be conducted as a telephone call if the participant has been discharged from the hospital or an in-person visit if the participant is still hospitalized).

For each participant, the total duration of the program is anticipated to be 4.5 months.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females ≥ 18 years of age and ≥ 40 kg at the time of providing informed consent.
2. Confirmed diagnosis of SARS-CoV-2 infection presenting as severe COVID-19 requiring hospitalization
3. Symptomatic, bilateral pulmonary infiltrates confirmed by CT or X-ray at Screening or within the 7 days prior to Screening
4. Severe pneumonia, acute lung injury, or ARDS requiring oxygen supplementation

Exclusion Criteria:

1. Confirmed diagnosis of SARS-CoV-2 infection presenting as mild to moderate COVID-19, even if the participant is hospitalized
2. Participant is not expected to survive more than 24 hours
3. Participant has an unresolved Neisseria meningitidis infection
4. Hypersensitivity to murine proteins or to one of the excipients of Soliris

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (12):
- United States (7):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Boston Medical Center, Boston, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
- France (5):
  - Hôpital Henri Mondor, Créteil
  - Hôpital Garches Raymond Poincaré, Garches
  - Hôpital de Bicêtre, Le Kremlin-Bicêtre
  - Hôpital Saint Louis, Paris
  - Hôpital Paul Brousse, Villejuif

REFERENCES:
- [Derived] Burwick RM, Dellapiana G, Newman RA, Smithson SD, Naqvi M, Williams J 3rd, Wong MS, Bautista M, Gaden A, Kazani SD, Dunn DA, Ma MH, Mitter S, Monteleone JPR, Ortiz SR, Ghandehari S, Merin N, Zakowski MI, Karumanchi SA. Complement blockade with eculizumab for treatment of severe Coronavirus Disease 2019 in pregnancy: A case series. Am J Reprod Immunol. 2022 Aug;88(2):e13559. doi: 10.1111/aji.13559. Epub 2022 May 12. PMID 35514201